CLINICAL TRIAL: NCT01144442
Title: WCC# 59: Pilot Study of Hyperthermic Intraperitoneal Chemotherapy Utilizing Carboplatin in First Recurrence
Brief Title: WCC# 59 Hyperthermic Intraperitoneal Chemotherapy Utilizing Carboplatin in First Recurrence Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Request
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS114; WCC# 59 (Other: Women's Cancer Center, University of Minnesota); 1003M78874 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-05-26; First posted 2010-06-15 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Carcinoma
Keywords: recurrent ovarian cancer; recurrent fallopian tube cancer; recurrent peritoneal carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Carboplatin; Sodium Chloride; Surgical Procedures, Operative; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPC Treatment (Experimental)
  Interventions: Drug: Hyperthermic intraperitoneal chemotherapy with Carboplatin; Other: Isotonic saline (perfusate); Procedure: Surgery; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Hyperthermic intraperitoneal chemotherapy with Carboplatin — Carboplatin at a dose of 1000mg/m^2 will be added to the perfusate once circulating levels reach 1000-1500cc/minute. The circulation of the chemotherapy impregnated perfusate will be performed for 90 minutes.
Other: Isotonic saline (perfusate) — The HIPC infusion will be performed with a closed abdomen technique. The perfusate will be isotonic saline heated to 40-42° Celsius.
  Other Names: saline
Procedure: Surgery — The abdominal incision will be performed in a vertical fashion extending from the supra-pubic region to around the umbilicus.
  If cytoreductive surgery is required, it will be performed at this time and proceed in standard approach.
Drug: Carboplatin — The scheduled systemic chemotherapy is paclitaxel 175mg/m2 and carboplatin AUC 6 every 3 weeks for 6 total cycles.
Drug: Paclitaxel — The scheduled systemic chemotherapy is paclitaxel 175mg/m2 and carboplatin AUC 6 every 3 weeks for 6 total cycles.
  Other Names: Taxol

SUMMARY:
This is an open-label, pilot study in patients with a diagnosis of recurrent ovarian, fallopian tube or primary peritoneal carcinoma who have undergone standard cytoreductive surgery following by adjuvant chemotherapy. It is expected that this first surgery was optimal - as defined as no residual tumor > or = 1 centimeter. Patient has clinical evidence of a first recurrence. The patient undergoes surgery and isotonic normal saline (perfusate) heated and administered into the abdomen, followed by hyperthermic intraperitoneal chemotherapy infusion (HIPC) administering carboplatin (chemotherapy). Six weeks after surgery patients will receive adjuvant chemotherapy with Paclitaxel and Carboplatin for 6 cycles.

DETAILED DESCRIPTION:
OBJECTIVES

* The primary objectives are

  * to determine the clinical response of hyperthermic intraperitoneal chemotherapy (HIPC) in patients at the time of first clinical recurrence of ovarian, fallopian tube, or primary peritoneal carcinoma
  * to determine the feasibility of delivering HIPC in a recurrent setting.
* Secondary objectives are

  * to determine disease free survival (DFS) and overall survival (OS),
  * to determine treatment related changes in quality of life (QOL)
  * to monitor the toxicities and complications associated with HIPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a histological diagnosis of primary ovarian, fallopian tube, or primary peritoneal carcinoma and have undergone chemotherapy according.
* Initial attempted cytoreductive surgery must have been performed by gynecologic oncologist with strict adherence to GOG surgical manual.
* End result of first surgery must have been optimal cytoreduction as defined as no residual tumor ≥ 1cm.
* Patients should have clinical evidence of first recurrence. Two fold elevations in CA125 or measurable tumor on CT scan constitute adequate evidence of recurrent disease.
* Patients with the following primary tumor epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, adenocarcinoma (non-specific) NOS, mixed epithelial carcinoma.
* Patients must have platin sensitive disease, defined as a recurrence occurring greater than 6 months from cessation of original treatment.
* Patients must have a performance status of 0, 1, 2.
* Patients must have adequate bone marrow function as defined by an absolute neutrophil count (ANC) ≥1500, platelet count ≥ 100,000, and a hemoglobin of greater than 10g/dl.
* Patients must have adequate renal function as defined by serum creatinine ≤ 1.5 mg/dl.
* Patients must have adequate hepatic function as defined by bilirubin ≤ 1.5 times normal levels, alkaline phosphatase and SGOT ≤ 3 times normal levels.
* Patients who have signed an Institutional Review Board (IRB) approved informed consent.
* Female patients 16-90 years of age.
* Patients must be deemed medically able to undergo a secondary surgical procedure.

Patient eligibility for systemic chemotherapy following HIPC:

* Patients must have successfully completed HIPC within 6 weeks of first prescribed intravenous carboplatin and taxane cycle.
* Patients must have a performance status of 0, 1, or 2.
* Patients must have adequate bone marrow function as defined as an ANC ≥ 1500, platelet count ≥ 100,000, and a hemoglobin of greater than 10g/dl.
* Patients must have adequate renal function as defined by serum creatinine ≤ 1.5 mg/dl.
* Patients must have adequate hepatic function as defined by bilirubin ≤ 1.5 times normal levels, alkaline phosphatase and SGOT ≤ 3 times normal levels.
* Patients who have signed an IRB approved informed consent.

Exclusion Criteria:

* Patients with known recurrent disease outside the abdominal cavity.
* Patients with low malignant tumor at primary diagnosis as determined by pathologic review.
* Patients with platin resistant disease as define as recurrence or progressive disease prior to 6 months from completion of primary therapy.
* Patients with any evidence of another malignancy within the last 5 years with the exception of non-melanoma skin cancer.
* Patients with evidence of concurrent septicemia, severe infection, renal failure, or acute hepatitis.
* Patients with history of grade 3 or greater gastrointestinal bleeding.
* Patients with a GOG performance score of 3 or 4.
* Patients deemed medically unable to tolerate the HIPC procedure by care giving physician.
* Patients with known allergy to platinum chemotherapy agents.
* Patients with equal to or greater than grade 2 neuropathy.

Ages: 16 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07-27 (Actual); Primary Completion 2013-09-25 (Actual); Study Completion 2015-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Argenta, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the Women's Health Clinic at the University of Minnesota. Recruitment occurred from September 2010 to April 2012.
Pre-assignment Details: Once subjects signed consent, they underwent cytoreductive surgery by a gynecologic oncologist with intent to resect all visible cancer. If subjects did not achieve optimal cytoreduction, they were ineligible.
Groups:
- HIPC Treatment: Patients treated with hyperthermic intraperitoneal chemotherapy at first recurrence of disease.
Period: Overall Study
Arm/Group | HIPC Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Customized [Median (Full Range); unit: years] | 56 (16.7) [47 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: We will summarize clinical response as the proportion of patients with complete response. Complete response will be defined as normalization of CA125. - After 6 cycles of Second Line Adjuvant Chemotherapy.
Time Frame: After 6 cycles of Paclitaxel & Carboplatin (Week 21 up to 27)
Measure: Number; unit: participants
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 10
participants | 10

2. Primary Outcome: Feasibility of HIPC in Recurrent Disease Setting
Description: We will determine feasibility based on the proportion of patients who complete 6 prescribed cycles of second line chemotherapy after undergoing the HIPC procedure.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 10
participants | 9

3. Secondary Outcome: Quality of Life Measurements
Description: The quality of life measurements (version 4 of the FACT-O questionnaire) will be summed over each subscale and overall and comparisons will be made using t-tests at distinct visits.
Time Frame: Baseline, 6 Weeks Post Surgery, Every 3 Weeks Up to Week 27
Population: Data was not collected due to the trial and all data collection processes being being terminated.
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Disease progression will be defined as time from surgery to first of either an increase in CA125 from post-treatment value (to a value greater than 100 or doubling of nadir CA125 levels) or new/increasing measurable disease by CT scan as defined by RECIST criteria, (secondary recurrence) or censored at date of last contact for patients still alive and who have no progressed or recurred (from date of surgery to disease progression).
Time Frame: Up to 5 Years (intended)
Population: Data was not collected due to the trial and all data collection processes being being terminated.
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as time from date of surgery to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: Up to 5 Years
Population: Data was not collected due to the trial and all data collection processes being being terminated.
Arm/Group | HIPC Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HIPC Treatment
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIPC Treatment (N=10)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Grade 3
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 4
Platelet count decreased (Investigations) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIPC Treatment (N=10)
Nausea (Gastrointestinal disorders) | 6 (6)
Ileus (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Transaminase abnormalties (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary weakness of this study is the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes